CLINICAL TRIAL: NCT05479903
Title: Clinical Study of the Relationship Between Different Interventions for Post-stroke Functional Impairment and Neurotrophic Factors
Brief Title: Study on the Correlation Between Neurotrophic Factors and the Condition of Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Lingcong Li, M.S. in Medicine, Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021kelunshen110
Record Dates: First submitted 2022-07-21; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Acupuncture Therapy; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- acupuncture stroke group (Experimental)
  Interventions: Procedure: acupuncture; Other: Conventional treatment
- sham acupuncture stroke group (Sham Comparator)
  Interventions: Other: Conventional treatment
- no acupuncture stroke group (Placebo Comparator)
  Interventions: Other: Conventional treatment
- acupuncture healthy group (Placebo Comparator)
  Interventions: Procedure: acupuncture
- computerized cognitive training group (Experimental)
  Interventions: Behavioral: computerized cognitive training system; Other: Conventional treatment
- tranditional cognitive training group (Placebo Comparator)
  Interventions: Behavioral: aerobic exercise; Other: Conventional treatment
- aerobics group (Experimental)
  Interventions: Behavioral: tranditional cognitive training; Other: Conventional treatment

INTERVENTIONS:
Procedure: acupuncture — Manual acupuncture or electro-acupuncture by experienced acupuncturists for patients
  Arms: acupuncture healthy group; acupuncture stroke group
Behavioral: computerized cognitive training system — One-on-one cognitive training by an experienced cognitive therapist, combined with an existing computerized cognitive training system
  Arms: computerized cognitive training group
Behavioral: aerobic exercise — Patients are trained by experienced physical therapists with the help of elastic bands and physical therapy devices
  Arms: tranditional cognitive training group
Behavioral: tranditional cognitive training — One-on-one cognitive training with an experienced cognitive therapist, combined with traditional cognitive training methods (e.g., balls, cards, counting, daily conversation, etc.)
  Arms: aerobics group
Other: Conventional treatment — Treatment of underlying disease and stroke according to guidelines, as well as necessary care and rehabilitation
  Arms: acupuncture stroke group; aerobics group; computerized cognitive training group; no acupuncture stroke group; sham acupuncture stroke group; tranditional cognitive training group

SUMMARY:
Stroke is currently the most common disabling disease, which often leads to impairment of sensory, motor, speech and psychological functions, resulting in a reduced quality of life for patients. Therefore, post-stroke functional rehabilitation, especially the rehabilitation of physical function and psychological condition, is particularly important for patients to rejoin society. Acupuncture can promote the functional recovery of patients and facilitate the rehabilitation of limb function, thus improving the quality of survival of post-stroke patients.

Neurotrophic factors are diverse, most of which are mainly derived from neuronal cells in the central nervous system and are involved in a variety of neurological functions such as cell growth, differentiation and plasticity, thus promoting recovery of multiple functions after stroke. Many studies have found that different interventions affect the prognosis of stroke patients differently, e.g., long-term acupuncture increases serum levels of brain-derived neurotrophic factor in stroke patients and also has better outcomes than controls in post-stroke neurological recovery and the development of post-stroke psychiatric disorders.

This study investigated the effects of different therapeutic measures on patients' functional recovery and neurotrophic factors by setting up a controlled and blinded trial design, which could not only provide clinical evidence for the effectiveness of relevant therapeutic measures, but also verify the clinical value of certain neurotrophic factors (e.g., predicting outcome, assessing condition, and preventing adverse events).

ELIGIBILITY:
Inclusion Criteria:

* Symptom recognition to admission ≤ 72 hours
* Clear imaging evidence
* Diagnosis of spontaneous cerebral hemorrhage by an immobilized physician according to relevant guidelines; pre-onset mRS score ≤ 1

Exclusion Criteria:

* This onset was caused by traumatic and violent factors
* History of previous intracranial surgery
* Previous cerebrovascular accident
* Previous speech disorders and limb movement disorders
* Participation in other trials in the last three months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
modified rankin scale | Change of the score of modified rankin scale from Baseline at 1 week after onset of disease
  The mrs (modified rankin scale) is a scale used to assess the patient's ability to care for himself/herself, which is composed of independent walking ability, self-perceived symptoms, and ability to control bowel and urine.Assessment results range from 0-6 points，a higher score means a worse ending
modified rankin scale | Change of the score of modified rankin scale from Baseline at 2 weeks after onset of disease
  The mrs (modified rankin scale) is a scale used to assess the patient's ability to care for himself/herself, which is composed of independent walking ability, self-perceived symptoms, and ability to control bowel and urine.Assessment results range from 0-6 points，a higher score means a worse ending
modified rankin scale | Change of the score of modified rankin scale from Baseline at 1 month after onset of disease
  The mrs (modified rankin scale) is a scale used to assess the patient's ability to care for himself/herself, which is composed of independent walking ability, self-perceived symptoms, and ability to control bowel and urine.Assessment results range from 0-6 points，a higher score means a worse ending
modified rankin scale | Change of the score of modified rankin scale from Baseline at 2 months after onset of disease
  The mrs (modified rankin scale) is a scale used to assess the patient's ability to care for himself/herself, which is composed of independent walking ability, self-perceived symptoms, and ability to control bowel and urine.Assessment results range from 0-6 points，a higher score means a worse ending
modified rankin scale | Change of the score of modified rankin scale from Baseline at 3 months after onset of disease
  The mrs (modified rankin scale) is a scale used to assess the patient's ability to care for himself/herself, which is composed of independent walking ability, self-perceived symptoms, and ability to control bowel and urine.Assessment results range from 0-6 points，a higher score means a worse ending

SECONDARY OUTCOMES:
Mini-mental State Examination | Change of the score of modified rankin scale from Baseline at 1 week, 2 weeks, 1 month, 2 months, 3 months after onset of disease
  The MMSE (Mini-mental State Examination) is a scale that assesses patients' cognition in terms of calculation, orientation, memory, and recall on a scale of 0-30, which is combined with the patient's level of education to yield results for different levels of cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Yongchuan Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No